CLINICAL TRIAL: NCT01731899
Title: Observational Study Evaluating the Efficacy and Tolerability of Agomelatine in the Treatment of Depressed Patients With Fibromyalgia
Brief Title: Agomelatine in Depressed Patients With Fibromyalgia
Status: Completed | Type: Observational
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Elena Pita Calandre, Professor, Universidad de Granada
Other Study IDs: AGO-2010
Record Dates: First submitted 2012-11-17; First posted 2012-11-22 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2014-05

CONDITIONS: Major Depression; Fibromyalgia
Keywords: major depression; fibromyalgia; agomelatine; Becks' Depression Inventory (BDI); Pittsburgh's Sleep Quality Index (PSQI)
MeSH Terms: conditions — Depressive Disorder, Major; Fibromyalgia | interventions — agomelatine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- agomelatine: patients diagnosed of fibromyalgia and concomitant major depression receiving agomelatine for this later disease
  Interventions: Drug: agomelatine

INTERVENTIONS:
Drug: agomelatine — Agomelatine 25 mg pills. Initial dose 25 mg at bedtime; can be increased up to 50 mg at bedtime; 12 weeks duration
  Other Names: Valdoxan

SUMMARY:
Depression and unrefreshed sleep are frequent in patients with fibromyalgia. Agomelatine is a new antidepressant with sleep-promoting properties. The objective of this study include the assessment of agomelatine therapy in patients with depression and fibromyalgia both on the severity of depressive symptomatology and sleep quality.

DETAILED DESCRIPTION:
One of the most frequent comorbidities of fibromyalgia is major depression. Agomelatine is a new antidepressant whose mechanims of action include both agonism at melatonin receptores and 5-HT2C blocking properties which, in addition to antidepressant efficacy, has shown sleep-improving properties. As unrefreshed sleep is a common symptom in fibromyalgia we hypothetized that agomelatine treatment of patients with concomitant depression and fibromyalgia could improve both depressive symtomatology and sleep quality. Thus, the objectives of the present study are the following:

* to assess the effectiveness and tolerability of agomelatine on the severity of depressive symptomatology in patients with fibromyalgia and concomitatnt depresssion
* to evaluate the effect of agomelatine treatment on sleep quality in these patients

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* diagnosed of fibromyalgia according to the American College of Rheumatology criteria
* diagnosed of major depression according to the DSM-IV criteria with a BDI-II score equal or higher tahn 20

Exclusion Criteria:

* other psychiastric concomitant illness
* pregnancy or lactation
* patients previously treated with agomelatine with little or no effect

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients suffering fibromyalgia and concomitant major depression
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2010-06; Primary Completion 2012-10 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
change, from baseline to endpoint, in the Beck's depression inventory score | 12 weeks

SECONDARY OUTCOMES:
change, from baseline to endpoint, in the Pittsburgh Sleep Quality Inventory | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Elena P Calandre, MD, Principal Investigator — Universidad de Granada
Locations (1):
- Instituto de Neurociencias, Granada, Granada, Spain

REFERENCES:
- [Result] Calandre EP, Slim M, Garcia-Leiva JM, Rodriguez-Lopez CM, Torres P, Rico-Villademoros F. Agomelatine for the treatment of patients with fibromyalgia and depressive symptomatology: an uncontrolled, 12-week, pilot study. Pharmacopsychiatry. 2014 Mar;47(2):67-72. doi: 10.1055/s-0033-1363659. Epub 2014 Feb 18. PMID 24549860